CLINICAL TRIAL: NCT02692586
Title: FlowTriever Pulmonary Embolectomy Clinical Study
Acronym: FLARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inari Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-001
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Results first posted 2021-04-29 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Embolism; Acute Pulmonary Embolism; Submassive Pulmonary Embolism; Massive Pulmonary Embolism
Keywords: Thromboembolism; Thrombectomy; Right Heart Strain; Submassive PE; Right Ventricle Dysfunction; Massive PE
MeSH Terms: conditions — Pulmonary Embolism; Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FlowTriever System (Experimental)
  Interventions: Device: FlowTriever System

INTERVENTIONS:
Device: FlowTriever System

SUMMARY:
Evaluate the safety and effectiveness of the FlowTriever System for use in the removal of emboli from the pulmonary arteries in the treatment of acute pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs, symptoms and presentation consistent with acute PE
* PE symptom duration ≤ 14 days
* CTA evidence of proximal PE
* RV/LV ratio ≥ 0.9 without syncope
* Systolic BP ≥ 90 mmHg
* Stable heart rate <130 BPM prior to procedure
* Patient deemed medically eligible for interventional procedure(s), per institutional guidelines and/or clinical judgment

Exclusion Criteria:

* Thrombolytic use within 30 days of baseline CTA
* Pulmonary hypertension with peak PAP > 70 mmHg by right heart catheterization
* Vasopressor requirement after fluids to keep pressure ≥ 90 mm Hg
* FiO2 requirement > 40% or > 6 LPM to keep oxygen saturation > 90%
* Hematocrit < 28% within 6 hours of index procedure
* Platelets < 100,000/µL
* Serum creatinine > 1.8 mg/dL
* INR > 3
* Major trauma ISS > 15
* Presence of intracardiac lead in right ventricle or atrium placed within 6 months
* Cardiovascular or pulmonary surgery within last 7 days
* Actively progressing cancer
* Known bleeding diathesis or coagulation disorder
* Left bundle branch block
* History of severe or chronic pulmonary arterial hypertension
* History of chronic left heart disease with left ventricular ejection fraction ≤ 30%
* History of uncompensated heart failure
* History of underlying lung disease that is oxygen-dependent
* History of chest irradiation
* History of Heparin-induced thrombocytopenia
* Any contraindication to systemic or therapeutic doses of heparin or anticoagulants
* Known anaphylactic reaction to radiographic contrast agents that cannot be pretreated
* Imaging evidence or other evidence that suggests the subject is not appropriate for mechanical thrombectomy intervention
* Life expectancy of < 90 days
* Female who is pregnant or nursing
* Current participation in another investigational drug or device treatment study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-04; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Rosenfield, MD, Study Chair — Massachusetts General Hospital; Victor Tapson, MD, Study Chair — Cedars-Sinai Medical Center
Locations (18):
- United States (18):
  - East Alabama Heart & Vascular, Auburn, Alabama
  - St. Vincent's, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Florida Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Ephraim McDowell Regional Medical Center, Danville, Kentucky
  - Baptist Health, Louisville, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - North Shore University Hospital, Manhasset, New York
  - Ohio State University, Columbus, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - UPMC Hamot, Erie, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
  - Charleston Area Medical Center, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- FlowTriever System: FlowTriever System
Period: Overall Study
Arm/Group | FlowTriever System
Started | 106
Completed | 103
Not Completed | 3
Not completed — Death from undiagnosed breast cancer through 30-day follow-up | 1
Not completed — Received adjunctive thrombolytics | 2

BASELINE CHARACTERISTICS:
Population: Measure Analysis Population Description: Measure Analysis Population Description: Study subjects with no thrombolytic agents administered during the index procedure (n = 104).
Arm/Group | FlowTriever System
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 103
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 17
  White | 86
  More than one race | 0
  Unknown or Not Reported | 0
Pre-procedural RV/LV ratio [Mean (Standard Deviation); unit: ratio] | 1.56 (0.34)

OUTCOME MEASURES:

1. Primary Outcome: Change in RV/LV Ratio
Description: Change in RV/LV ratio from baseline to 48 hours
Time Frame: Baseline to 48 hours
Population: Patients with symptomatic, computed tomography-documented PE and RV/LV ratios ≥ 0.9 treated with the FlowTriever System that were not administered thrombolytic agents during the index procedure (n = 104)
Measure: Mean (Standard Error); unit: RV/LV ratio
Groups:
- FlowTriever System: Patients treated with the FlowTriever System
Arm/Group | FlowTriever System
Number analyzed (Participants) | 104
RV/LV ratio | 0.38 (0.03)
Statistical Analysis 1: Comparison: FlowTriever System; Test type: Superiority — To detect an RV/LV ratio change > 0.12 with a power of 80% at one-sided alpha = 0.025, the necessary sample size was calculated to be ≥ 52, 31, or 21 patients (to detect RV/LV ratio changes of 0.20, 0.225, or 0.25, respectively); p < 0.0001, t-test, 1 sided

2. Primary Outcome: Number of Participants With Major Adverse Events
Description: Device-related death, major bleeding, and treatment related AEs
Time Frame: Within 48 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever System
Number analyzed (Participants) | 104
Participants
  Participants experiencing MAEs | 4
  Participants not experiencing MAEs | 100
Statistical Analysis 1: Comparison: FlowTriever System; Test type: Superiority — The hypothesized composite MAE rate was expected to be about 13%. The necessary sample size to detect a difference from an expected MAE rate of 13% with 80% power was calculated to be 103 patients (with a one-sided p value = 0.05); p < 0.0001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 30 +/- 3 days
Arm/Group | FlowTriever System
All-Cause Mortality (participants affected / at risk) | 1/106
Serious Adverse Events (participants affected / at risk) | 14/106
Other Adverse Events (participants affected / at risk) | 0/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FlowTriever System (N=106)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Catheter site hematoma (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Acute respiratory failure (Metabolism and nutrition disorders) | 1 (1)
Respiratory failure (Metabolism and nutrition disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT02692586/Prot_SAP_000.pdf